CLINICAL TRIAL: NCT03211572
Title: Evaluating Multiparameter Gene Testing as a Predictor of Short Term Endocrine Therapy Response in Hormone Receptor Positive Breast Cancers: The EMPOwER Study
Brief Title: The EMPOwER Study Evaluating Multiparameter Gene Testing as a Predictor of Short Term Endocrine Therapy Response in Hormone Receptor Positive Breast Cancers
Acronym: OTT 17-01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20170345-01h
Record Dates: First submitted 2017-07-05; First posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer
Keywords: breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Anastrozole

STUDY DESIGN:
Intervention Model Description: The clinical trial will be a prospective, two-strata, non-blinded, single institution Health Canada approved window of opportunity trial with 2 weeks of pre-surgical endocrine therapy using either anastrozole or tamoxifen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endocrine Therapy (Experimental): Anastrozole 1 mg (postmenopausal) or tamoxifen 20mg (premenopausal) are to be taken orally each evening and would be started exactly 2 weeks prior to their surgery.
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen — Participants will take endocrine therapy for 2 weeks prior to surgery.
  Other Names: Anastrozole

SUMMARY:
Evaluating Multiparameter Gene Testing as a Predictor of Short Term Endocrine Therapy Response in Hormone Receptor Positive Breast Cancers

DETAILED DESCRIPTION:
The clinical trial will be a prospective, two strata, non-blinded, single institution, Health Canada approved, Window of Opportunity trial with 2 weeks of pre-surgical endocrine therapy using either anastrozole or tamoxifen. Tissue from the initial biopsy and from surgery will be sent for Ki67 analysis using the NanoString® Assay.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with histologically confirmed newly diagnosed operable ER+, Her2 negative invasive carcinoma on diagnostic core biopsy that has a radiographic size ≥ 1.5 cm
* Histology has to be ductal, lobular or mixed
* Surgery date planned in the next 2-6 weeks
* Negative pregnancy test if of child baring potential
* Post-menopausal status verified by FSH and Estradiol (with 6 months of amenorrhea)

Exclusion Criteria:

* Previous treatment with endocrine therapy, chemotherapy or chest wall radiation within last 6 months
* Known metastatic or recurrent breast cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Endocrine Therapy response | at one year
  Introduction and validation of the use of NanoString® technology and a development of a custom gene codeset predictive of endocrine therapy response into the window setting as a more robust and reliable method of biomarker assessment as compared to Ki67.

SECONDARY OUTCOMES:
Biomarker Predictive value | at one year
  Window of Opportunity clinical trial design as a means to evaluate the predictive value of potential biomarkers or biomarker-based tools.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Arnaout, Dr., Principal Investigator — The Ottawa Hospital

IPD SHARING:
Plan to Share IPD: No